CLINICAL TRIAL: NCT03122353
Title: A Randomized, Double-Blind Study Comparing TOLMAR Calcipotriene and Betamethasone Suspension to Reference Listed Drug in the Treatment of Scalp Psoriasis
Brief Title: BE Study of Calcipotriene Hydrate and Betamethasone Dipropionate Topical Suspension in the Treatment of Scalp Psoriasis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tolmar Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TOL2708C
Record Dates: First submitted 2017-04-06; First posted 2017-04-20 (Actual); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Scalp Psoriasis
MeSH Terms: interventions — calcipotriene; Betamethasone; betamethasone dipropionate, calcipotriol drug combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Calcipotriene Hydrate and Betamethasone (Experimental): Calcipotriene hydrate and betamethasone dipropionate topical suspension 0.005%/0.064%
  Interventions: Drug: Calcipotriene and betamethasone suspension
- Taclonex (Active Comparator): Calcipotriene hydrate and betamethasone dipropionate topical suspension 0.005%/0.064%
  Interventions: Drug: Taclonex
- Placebo (Placebo Comparator): Topical suspension without active ingredient
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Calcipotriene and betamethasone suspension — Calcipotriene hydrate and betamethasone dipropionate topical suspension 0.005%/0.064%
  Other Names: Calcipotriene, betamethasone
  Arms: Calcipotriene Hydrate and Betamethasone
Drug: Taclonex — Calcipotriene hydrate and betamethasone dipropionate topical suspension 0.005%/0.064%
  Other Names: Calcipotriene, betamethasone
  Arms: Taclonex
Drug: Placebo — vehicle used as placebo
  Other Names: Vehicle
  Arms: Placebo

SUMMARY:
This study will be conducted to evaluate the therapeutic bioequivalence of a TEST formulation of calcipotriene hydrate and betamethasone dipropionate topical suspension 0.005%/0.064% to the RLD.

DETAILED DESCRIPTION:
Randomized, Double-Blind, Placebo-Controlled, Multiple-Site, Parallel Design, Bioequivalence with Clinical Endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant, non-lactating female, at least 18 years of age.
* Female subjects of childbearing potential (excluding women who are or premenarchal, surgically sterilized or postmenopausal for at least 2 years).
* A clinical diagnosis of stable (at least 6 months) scalp psoriasis involving at least 10% of the scalp and clinical signs of psoriasis vulgaris on trunk and/or limbs.
* Scalp psoriasis consistent with at least moderate disease severity (grade ≥ 3) using the Physician's Global Assessment (PGA) of disease severity.
* Plaque elevation of at least moderate severity (grade ≥ 3) at the scalp target lesion site using the Psoriasis Area Severity Index (PASI). The most severe lesion at Baseline will be identified as the scalp target lesion.
* Agree to stop use of all other topical or systemic antipsoriatic treatments, corticosteroids, immunosuppressive drugs, calcium supplements and Vitamin D supplements or Vitamin D analogs at a dose > 400 IU/day during the study.
* Currently in general good health and free from any clinically significant disease, other than scalp psoriasis and psoriasis vulgaris, that may interfere with the study evaluations.
* Willing and able to understand and comply with the requirements of the study, apply IP as instructed, attend required study visits, comply with study prohibitions, and be able to complete the study.

Exclusion Criteria:

* Current diagnosis of unstable forms of psoriasis including guttate, erythrodermic, exfoliative or pustular psoriasis.
* Other inflammatory skin disease in the scalp that may confound the evaluation of the scalp psoriasis (eg, atopic dermatitis, contact dermatitis, tinea capitis).
* History of hypersensitivity to any component of TEST or RLD.
* Current or past history of hypercalcemia, hypercalciuria, vitamin D toxicity, severe renal insufficiency, or hepatic disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 699 (Actual)
Dates: Start 2017-04-11 (Actual); Primary Completion 2017-11-15 (Actual); Study Completion 2017-11-15 (Actual)

PRIMARY OUTCOMES:
Psoriasis Area Severity Index (PASI) | at Day 1, Day 28
  To evaluate the change in clinical outcome of patients exposed to Calcipotriene hydrate and betamethasone dipropionate topical suspension 0.005%/0.064%, Taclonex and Vehicle for scalp psoriasis. From baseline to end of study.
Physician Global Assessment (PGA) | at Day 1, Day 28
  To evaluate the change in global severity of skin of patients exposed to Calcipotriene hydrate and betamethasone dipropionate topical suspension 0.005%/0.064%, Taclonex, and Vehicle for scalp psoriasis. From baseline to end of study.
Body Surface Area (BSA) | at Day 1
  To evaluate the total body area of skin affected by psoriasis.
Adverse Events and Serious Adverse Events | at Day 28
  Risk for adverse events and serious adverse events for exposed to Calcipotriene hydrate and betamethasone dipropionate topical suspension 0.005%/0.064%, Taclonex and Vehicle for scalp psoriasis

CONTACTS AND LOCATIONS:
Overall Officials: Jim Joffrion, Study Director — Catawba Research
Locations (34):
- United States (34):
  - Site 17, Hot Springs, Arkansas
  - Site 29, Fremont, California
  - Site 12, Los Angeles, California
  - Site 18, Sherman Oaks, California
  - Site 34, Denver, Colorado
  - Site 20, Boca Raton, Florida
  - Site 01, Brandon, Florida
  - Site 25, Coral Gables, Florida
  - Site 11, Hialeah, Florida
  - Site 26, Miami, Florida
  - Site 04, Miami, Florida
  - Site 05, Miramar, Florida
  - Site 02, Tampa, Florida
  - Site 03, Tampa, Florida
  - Site 23, Winter Park, Florida
  - Site 16, Plainfield, Indiana
  - Site 19, Olathe, Kansas
  - Site 33, Lake Charles, Louisiana
  - Site 27, Saint Joseph, Missouri
  - Site 14, Las Vegas, Nevada
  - Site 09, High Point, North Carolina
  - Site 28, Hazleton, Pennsylvania
  - Site 24, Upper Saint Clair, Pennsylvania
  - Site 32, Johnston, Rhode Island
  - Site 07, Anderson, South Carolina
  - Site 35, Mt. Pleasant, South Carolina
  - Site 21, Austin, Texas
  - Site 06, Dallas, Texas
  - Site 30, El Paso, Texas
  - Site 08, Murphy, Texas
  - Site 15, San Antonio, Texas
  - Site 31, San Antonio, Texas
  - Site 10, Salt Lake City, Utah
  - Site 22, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No